CLINICAL TRIAL: NCT01307228
Title: Effects of an Evidence Service on Health System Policymakers' Use of Research Evidence
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient participants recruited for the trial
Sponsor: McMaster University (Other)
Collaborators: Ontario Ministry of Health and Long Term Care (Other Government)
Responsible Party: Principal Investigator, John Lavis, Professor, Department of Health Evidence and Impact, McMaster University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: HHS/FHS REB 10-267
Record Dates: First submitted 2011-02-28; First posted 2011-03-02 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Use of Research Evidence
Keywords: Knowledge translation; Policymakers; Health systems

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Full-serve evidence service (Experimental): The "full-serve" evidence service consists of:
  1. database (Health Systems Evidence) access;
  2. monthly e-mail alerts; and
  3. full-text article availability.
  Interventions: Other: Health Systems Evidence
- Self-serve evidence service (Active Comparator): Participants allocated to the "self-serve" evidence service will receive only database access, which is already publicly available at www.healthsystemsevidence.org
  Interventions: Other: Health Systems Evidence

INTERVENTIONS:
Other: Health Systems Evidence — Health Systems Evidence (HSE) contains over 1400 research syntheses about governance, financial and delivery arrangements within health systems and about implementation strategies relevant to health systems. The syntheses have been: 1) categorized by topic, type of synthesis, and type of question addressed; 2) coded by the last year in which searches for studies were conducted and by the countries in which included studies were conducted; 3) rated for quality; and 4) linked to publicly available user-friendly summaries, scientific abstracts, and full-text reviews. We identified systematic reviews in HSE that are not accessible to study participants and developed a mechanism to reimburse publishers for full-text downloads of these reviews.

SUMMARY:
The investigators have developed an online database called 'Health Systems Evidence,' which contains synthesized research evidence and additional details about this evidence that can make it easier for health system policymakers to use the included research evidence. The investigators have also developed an e-mail alerting service that brings to the attention of health system policymakers any new additions to Health Systems Evidence. This study will evaluate whether a "full-serve" version of Health Systems Evidence increases the use of research evidence by policy analysts and advisors in the Ontario government as compared to a "self-serve" version. The "full-serve" version comprises: 1) access to Health Systems Evidence; 2) monthly e-mail alerts about new additions to Health Systems Evidence; and 3) access to full-text articles that are cited in Health Systems Evidence. The "self-serve" version only provides access to Health Systems Evidence. The investigators will also interview study participants to obtain feedback about Health Systems Evidence, including how helpful it was in their work, why it was helpful (or not helpful), what aspects were most and least helpful and why, and recommendations for improving it.

DETAILED DESCRIPTION:
Background Health system policymakers need timely access to synthesized research evidence to inform the policymaking process. No efforts to address this need have been evaluated using an experimental quantitative design. The investigators developed an evidence service that draws inputs from Health Systems Evidence, which is a database of policy relevant systematic reviews. The reviews have been: 1) categorized by topic and type of review; 2) coded by the last year searches for studies were conducted and by the countries in which included studies were conducted; 3) rated for quality; and 4) linked to available user-friendly summaries, scientific abstracts, and full-text reports. The goal is to evaluate whether a "full-serve" evidence service increases the use of synthesized research evidence by policy analysts and advisors in the Ontario Ministry of Health and Long-Term Care (MOHLTC) as compared to a "self-serve" evidence service.

Methods/design: The investigators will conduct a two-arm randomized controlled trial (RCT), along with a follow-up qualitative process study in order to explore the findings in greater depth. For the RCT, all policy analysts and policy advisors (n=168) in a single division of the MOHLTC will be invited to participate. Using a stratified randomized design, participants will be randomized to receive either the "full-serve" evidence service (database access, monthly e-mail alerts, and full-text article availability) or the "self-serve" evidence service (database access only). The trial duration will be ten months (two-month baseline period, six-month intervention period, and two month cross-over period). The primary outcome will be the mean number of site visits/month/user between baseline and the end of the intervention period. The secondary outcome will be participants' intention to use research evidence. For the qualitative study, 15 participants from each trial arm (n=30) will be purposively sampled. One-on-one semi-structured interviews will be conducted by telephone on their views about and their experiences with the evidence service they received, how helpful it was in their work, why it was helpful (or not helpful), what aspects were most and least helpful and why, and recommendations for next steps.

ELIGIBILITY:
Inclusion Criteria:

* All policy analysts and policy advisors from one purposively selected division of one Canadian provincial Ministry of Health.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2011-04 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
number of logins/month/participant | 10 months
  The investigators will track utilization of the evidence service by calculating the mean number of logins/month/participant

SECONDARY OUTCOMES:
Intention to use research evidence | Baseline and follow-up (after delivery of 6-month intervention)
  The investigators will use the theory of planned behaviour to measure participants' intention to use research evidence. Using a manual designed to construct measures based on the theory, colleagues have developed and sought preliminary feedback on a data-collection instrument by first assessing face validity through interviews with key informants and then pilot testing it with 28 policymakers and researchers who completed it after participating in a knowledge translation intervention. In addition, colleagues found the data-collection instrument to have moderate test-retest reliability.

CONTACTS AND LOCATIONS:
Overall Officials: John N Lavis, MD, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster Health Forum Impact Lab, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Not applicable - trial was terminated due to insufficient enrollment and no data was collected.

REFERENCES:
- [Derived] Lavis JN, Wilson MG, Grimshaw JM, Haynes RB, Hanna S, Raina P, Gruen R, Ouimet M. Effects of an evidence service on health-system policy makers' use of research evidence: a protocol for a randomised controlled trial. Implement Sci. 2011 May 27;6:51. doi: 10.1186/1748-5908-6-51. PMID 21619621